CLINICAL TRIAL: NCT05693363
Title: Perioperative Specimen Imaging Using High-resolution 18F-FDG-PET-CT During Thoracic Surgery: a Pilot Study
Acronym: ThorPET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: XEOS Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ONZ-2023-0105
Record Dates: First submitted 2023-01-11; First posted 2023-01-23 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Lung Neoplasms; PET-CT Specimen Imager
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-FDG AURA10 Specimen Imager (Experimental): * Intravenous injection of radiotracer (18F-FDG) (study-specific)
  * Thoracic surgery (standard-of-care; not study-specific)
  * High-resolution specimen imaging using the AURA10 PET-CT specimen imager (study-specific)
  * Postoperative histopathological analysis of specimen (standard-of-care)
  Interventions: Device: AURA10 Specimen Imager

INTERVENTIONS:
Device: AURA10 Specimen Imager — High-resolution specimen imaging using the AURA10 PET-CT specimen imager during thoracic surgery.

SUMMARY:
In this pilot study the investigators propose the intraoperative use of a high-resolution PET-CT imaging system which can assess resection margins and lymph node status in the operating room. This will allow for a faster and stepwise assessment (estimated to be under 10 minutes per specimen), enabling the surgeon to decide on subsequent surgical steps after each previous assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older.
* Patient with suspected or confirmed lung malignancies
* Patient is indicated to undergo thoracic surgery.
* Patient is estimated to be compliant for study participation by the investigator.
* Patient has freely given his/her informed consent to participate in this study.

Exclusion Criteria:

* Patient has general or local contra-indications for thoracic surgery.
* Patient has active infection.
* Blood glucose level over 200 mg/dL on the day of surgery.
* Pregnancy or lactation.
* Patient participated in other clinical studies with radiation exposure of more than 1 mSv in the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Perioperative success in imaging utilizing AURA10 PET-CT Specimen Imager | Perioperative
  A measure of perioperative success in imaging 18F-FDG- uptake in resected specimens obtained during thoracic surgery utilizing a high-resolution PET-CT-scanner.

SECONDARY OUTCOMES:
Sensitivity and specificity of high-resolution 18F-FDG-PET-CT of resected mediastinal or thoracic lymph nodes in terms of nodal staging. | Perioperative
Sensitivity and specificity of high-resolution 18F-FDG-PET-CT of resected lung tumors in terms of bronchial margin assessment. | Perioperative
Sensitivity and specificity of high-resolution 18F-FDG-PET-CT of resected lung tumors in terms of lung parenchyma margin assessment | Perioperative
Correlation between 18F-FDG uptake in the resected specimens and histopathological characteristics of the tumor, such as the type, grade, or stage of the tumor. | Perioperative
Measure signal-to-noise ratio on post-processed PET-CT specimen images. | Perioperative
Comparison of lesion dimensions (e.g. delineation based on percentage of SUVmax, tumor-to-background ratios based on SUVpeak). | Perioperative
Occupational radiation exposure (µSv) to the staff in the operating room related to this study. | Perioperative
Correlation of high-resolution 18F-FDG-PET-CT images of lamellas of the resected specimen with histopathological whole-slide images. | Perioperative

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goker M, Marcinkowski R, Van Bockstal M, Keereman V, Van Holen R, Van Dorpe J, Vandenberghe S, Brans B, Depypere H, Van den Broecke R. 18F-FDG micro-PET/CT for intra-operative margin assessment during breast-conserving surgery. Acta Chir Belg. 2020 Oct;120(5):366-374. doi: 10.1080/00015458.2020.1774163. Epub 2020 Jun 15. PMID 32452298
- [Background] Piron S, De Man K, Van Laeken N, D'Asseler Y, Bacher K, Kersemans K, Ost P, Decaestecker K, Deseyne P, Fonteyne V, Lumen N, Achten E, Brans B, De Vos F. Radiation Dosimetry and Biodistribution of 18F-PSMA-11 for PET Imaging of Prostate Cancer. J Nucl Med. 2019 Dec;60(12):1736-1742. doi: 10.2967/jnumed.118.225250. Epub 2019 Apr 26. PMID 31028165
- See also: J. Ferlay, M. Ervik, F. Lam, M. Colombet, L. Mery, and M. Piñeros, "Global Cancer Observatory: Cancer Today. Lyon: International Agency for Research on Cancer." 2020 — https://gco.iarc.fr/today